CLINICAL TRIAL: NCT00793364
Title: Effect of Plant Stanol Ester-Containing Spread Based on Extra Virgin Olive Oil on Estimated Cardiovascular Risk, and Lipid-Inflammatory-Haemostatic Factors in Comparison to Mediterranean Diet: A Randomized, Placebo-Controlled Trial.
Brief Title: Effect of Plant Stanol Ester-Containing Spread on Estimated Cardiovascular Risk in Comparison to Mediterranean Diet
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hellenic Atherosclerosis Society (Other)
Collaborators: Minerva SA (Industry)
Responsible Party: Vasilios G. Athyros, MD / Professor / Primary investigator, Hippocration Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MINERVA 01; 171108
Record Dates: First submitted 2008-11-17; First posted 2008-11-19 (Estimated); Last update posted 2009-05-28 (Estimated); Status verified 2009-05

CONDITIONS: Hypercholesterolemia
Keywords: Cholesterol, stanol-ester, mediterranean diet, cardiac risk
MeSH Terms: conditions — Hypercholesterolemia | interventions — Dietary Supplements; Diet, Mediterranean

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Stanol ester (Active Comparator): Stanol-ester administration group
  Interventions: Dietary Supplement: Stanol ester spread
- Placebo spread (Placebo Comparator): Placebo spread group
  Interventions: Dietary Supplement: Placebo spread
- Mediterranean diet group (Other): Mediterranean diet group
  Interventions: Dietary Supplement: Mediterranean Diet

INTERVENTIONS:
Dietary Supplement: Stanol ester spread — Stanol ester spread 20 g every day
  Other Names: Dietary Supplement
  Arms: Stanol ester
Dietary Supplement: Placebo spread — Placebo spread 20 g every day
  Other Names: Dietary Supplement
  Arms: Placebo spread
Dietary Supplement: Mediterranean Diet — Mediterranean Diet every day
  Other Names: Dietary Supplement
  Arms: Mediterranean diet group

SUMMARY:
Since it is very difficult to have the real thing (Mediterranean diet) we need to find an alternative to reduce cardiovascular disease (CVD) risk in subjects with moderate hypercholesterolaemia (a major CVD risk factor) living in western countries. Therefore, this proposed study is designed to assess if giving olive oil supplements, with or without stanol ester, is equivalent to following a Mediterranean diet. Furthermore, the stanol-olive oil combination may prove to be superior to olive oil alone.

DETAILED DESCRIPTION:
Design: Randomised, double blind, placebo controlled study Number of participants: 150 (3 groups with 50 subjects each). Intervention: One group will be assigned to stanol ester spread (2 g/day) based on olive oil, another on spread with olive oil containing placebo stanol ester (in identical containers with the stanol ester spread). In the third group, a structured effort will be made to improve adherence to Mediterranean diet by at least 2 points in a 10-level scale. Adherence to the Mediterranean diet will be improved by a dietician with detailed explanation of the composition of the diet, preparation of several week specific programs according to dietary preferences of the specific subject. Dietician interviews with a 5 day questionnaire on consumed foods will establish the degree of adherence to Mediterranean diet.

Duration: 16 weeks (4 weeks of lifestyle advice and 12 weeks of treatment).

Prespecified analyses:

1. Postmenopausal women vs women with child bearing potential.
2. Older (>65 years of age) vs younger subjects,
3. Subjects with impaired fasting glucose levels.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects over 45 years of age with mild hypercholesterolaemia (TC levels: 200 mg/dl - 230 mg/dl)

Exclusion Criteria:

Subjects with

* Established CVD (coronary heart disease, peripheral arterial disease, aortic aneurysm, or symptomatic carotid artery disease) or T2DM
* Chronic diseases (including liver diseases)
* Pregnancy
* Malignancies
* Unwillingness to participate

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2008-11; Primary Completion 2009-03 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Primary endpoint: Change from baseline in cardiovascular (CVD) risk as assessed by the PROCAM and Framingham risk engines. | three months

SECONDARY OUTCOMES:
Change from baseline in major CVD risk factors [TC, LDL-C, HDL-C, TG, apoB], in an inflammatory marker [C-reactive protein], in hemostatic parameters (PAI-I, fibrinogen), liver function tests at the end of the study vs baseline. | three months

CONTACTS AND LOCATIONS:
Overall Officials: Vasilios G Athyros, MD, Principal Investigator — Hippocration Hospital
Locations (1):
- Aristotelian University, Hippocration Hospital, Thessaloniki, Greece

REFERENCES:
- [Result] Nguyen TT, Dale LC, von Bergmann K, Croghan IT. Cholesterol-lowering effect of stanol ester in a US population of mildly hypercholesterolemic men and women: a randomized controlled trial. Mayo Clin Proc. 1999 Dec;74(12):1198-206. doi: 10.4065/74.12.1198. PMID 10593347
- [Derived] Athyros VG, Kakafika AI, Papageorgiou AA, Tziomalos K, Peletidou A, Vosikis C, Karagiannis A, Mikhailidis DP. Effect of a plant stanol ester-containing spread, placebo spread, or Mediterranean diet on estimated cardiovascular risk and lipid, inflammatory and haemostatic factors. Nutr Metab Cardiovasc Dis. 2011 Mar;21(3):213-21. doi: 10.1016/j.numecd.2009.08.014. Epub 2009 Nov 25. PMID 19939653